CLINICAL TRIAL: NCT01558622
Title: Intraoperative Use of Dexketoprofen Trometamol, Tramadol Hcl, Pethidine Hcl and Their Combinations for Postoperative Pain Management in Laparoscopic Nissen Fundoplication
Brief Title: Intraoperative Use of Dexketoprofen Trometamol, Pethidine Hcl, Tramadol Hcl and Their Combinations for Postoperative Pain Management in Laparoscopic Nissen Fundoplication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kavaklıdere Umut Hospital (Other)
Responsible Party: Principal Investigator, GOKHAN GOKMEN, Anesthesiologist, MD, Kavaklıdere Umut Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KVDU 0001 GG
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Laparoscopic Nissen Fundoplication
Keywords: postoperative analgesia; dexketoprofen trometamol; tramadol hydrochloride; pethidine; laparoscopic Nissen fundoplication
MeSH Terms: interventions — dexketoprofen trometamol; Tramadol; Meperidine; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- dexketoprofen trometamol (Placebo Comparator): Dexketoprofen trometamol is a water-soluble salt of the dextrorotatory enantiomer of the nonsteroidal anti-inflammatory drug (NSAID) ketoprofen.
  Interventions: Drug: dexketoprofen trometamol
- tramadol hydrochloride (Placebo Comparator): Tramadol Hydrochloride is a well-known centrally acting opioid pain killer.
  Interventions: Drug: tramadol hydrochloride
- pethidine hydrochloride (Placebo Comparator): Pethidine is a synthetic opioid analgesic which produces a pattern of effects similar to morphine the standard against which opioid analgesics are compared.
  Interventions: Drug: pethidine hydrochloride
- dexketoprofen trometamol + tramadol hydrochloride (Placebo Comparator)
  Interventions: Drug: dexketoprofen trometamol + tramadol hydrochloride
- dexketoprofen trometamol + pethidine hydrochloride (Placebo Comparator)
  Interventions: Drug: dexketoprofen trometamol + pethidine hydrochloride
- vitamin c (Placebo Comparator)
  Interventions: Drug: vitamin c

INTERVENTIONS:
Drug: dexketoprofen trometamol — 50mg intravenous infusion
  Arms: dexketoprofen trometamol
Drug: tramadol hydrochloride — 100mg intravenous infusion
  Arms: tramadol hydrochloride
Drug: pethidine hydrochloride — 50mg intravenous infusion
  Arms: pethidine hydrochloride
Drug: dexketoprofen trometamol + tramadol hydrochloride — intravenous infusion of 50mg dexketoprofen trometamol + 100mg tramadol hydrochloride
  Arms: dexketoprofen trometamol + tramadol hydrochloride
Drug: dexketoprofen trometamol + pethidine hydrochloride — intravenous infusion of 50mg dexketoprofen trometamol + 50mg pethidine hydrochloride
  Arms: dexketoprofen trometamol + pethidine hydrochloride
Drug: vitamin c — 500mg intravenous infusion
  Arms: vitamin c

SUMMARY:
The purpose of this study is to evaluate the analgesic effects of dexketoprofen trometamol, tramadol hydrochloride, pethidine hydrochloride and their combinations in laparoscopic Nissen fundoplication.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old ASA I-II patients
* Clinical diagnosis of gastroesophageal reflux patients

Exclusion Criteria:

* Allergic reactions to NSAIDs or opioid analgesics
* Body mass index exceeding 35
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Allergic reactions to NSAIDs or opioid analgesics, body mass index exceeding 35 | postoperative 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: GOKHAN GOKMEN, Specialist, Principal Investigator
Locations (1):
- Kavaklidere Umut Hospital, Ankara, Turkey (Türkiye)